CLINICAL TRIAL: NCT05126784
Title: A Randomized, Double-blind, Single-dose, Parallel-group Design, 2 Arm Study Comparing the Pharmacokinetic, Pharmacodynamic, Safety, Tolerability, and Immunogenicity Profiles of AVT03 and Prolia® in Healthy Male Subjects
Brief Title: AVT03 With Prolia in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alvotech Swiss AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: AVT03-GL-P01
Record Dates: First submitted 2021-11-01; First posted 2021-11-19 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Healthy Male Subjects
Keywords: Denosumab; Healthy Volunteers
MeSH Terms: interventions — Denosumab

STUDY DESIGN:
Intervention Model Description: Arm 1: AVT03 Arm 2: US-Prolia
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double Blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- AVT03 Arm (Experimental): AVT03 (denosumab) is the proposed biosimilar for Prolia (denosumab). Subjects in this arm will receive a single 60mg dose of AVT03 (denosumab) as a subcutaneous injection.
  Interventions: Biological: AVT03
- Prolia Arm (Active Comparator): Prolia(denosumab) is the proposed comparator for AVT03 (denosumab). Subjects in this arm will receive a single 60mg dose of Prolia (denosumab) as a subcutaneous injection.
  Interventions: Biological: Prolia

INTERVENTIONS:
Biological: AVT03 — AVT03 (biosimilar to denosumab) will be given as single subcutaneous injection
  Other Names: AVT03, Biosimilar Denosumab
  Arms: AVT03 Arm
Biological: Prolia — Prolia (denosumab) will be given as single subcutaneous injection
  Other Names: Denosumab
  Arms: Prolia Arm

SUMMARY:
This study has been designed as a randomized, double-blind, single-dose, parallel-group study in healthy adult male subjects 28 years to 55 years old. The study will assess the PK, PD, safety, tolerability and immunogenicity of AVT03 compared to Prolia when administered as a single SC dose.

DETAILED DESCRIPTION:
The study will consist of a 4 week screening period, a 252 day (36 weeks) treatment and assessment period, and an End of Study (EOS) visit on week 36 on Day 252. Subjects will undertake a screening visit between Day -28 and Day -1 to determine their eligibility for the study. On Day 1, eligible subjects will be randomized and will receive a single dose of AVT03 or Prolia as subcutaneous injection.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects who are 28 to 55 years old, inclusive
* Have a body weight of 50.0 to 90.0 kg (inclusive) and body mass index (BMI) of 17.0 to 32.0 kg/m2 (inclusive)at Screening and Day -1
* Medical history without evidence of a clinically significant disorder, condition, or disease that, in the opinion of the Investigator, would pose a risk to subject safety

Exclusion Criteria:

* Any evidence of clinically relevant pathology, especially prior diagnosis of bone disease, or any uncontrolled condition that will affect bone metabolism (such as, but not limited to osteoporosis, osteogenesis imperfecta, hyperparathyroidism, hyperthyroidism, hypothyroidism, osteomalacia, rheumatoid arthritis, psoriatic arthritis, ankylosing spondylitis, current flare-up of osteoarthritis and/or gout, active malignancy, renal disease, Paget's disease of the bone, recent bone fracture [within 6 months], and malabsorption syndrome)
* Have osteonecrosis of the jaw (ONJ) or risk factors for ONJ such as invasive dental procedures (eg, tooth extraction, dental implants, oral surgery) within 6 months prior to Day 1 or intend to undergo such procedures during the study period, poor oral hygiene, periodontal, and/or pre existing dental disease
* Have bone fractures within 6 months prior to Day -1.
* Have a history of immunodeficiency
* Those with skin allergies, or are susceptible to autoinflammatory skin disorders, or prone to the development of allergic skin inflammation
* Abnormal serum calcium: current hypocalcemia or hypercalcemia at Screening. Serum calcium levels must be within reference ranges.
* Known vitamin D deficiency

Ages: 28 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 209 (Actual)
Dates: Start 2022-06-29 (Actual); Primary Completion 2023-10-16 (Actual); Study Completion 2023-10-16 (Actual)

PRIMARY OUTCOMES:
Area under the serum concentration-time curve (AUC0-last) from day 0 to day 252 | Day 1(week 1) to Day 252 (week 36)
  Venous blood samples will be collected for measurement of Area under serum concentration-time curve (AUC 0-t) AVT03 and Prolia
Area under the serum concentration-time curve (AUC0-inf) from day 0 to day 252 | Time Frame: Day 1(week 1) to Day 252 (week 36)]
  Venous blood samples will be collected for measurement of CTX-1 serum biomarker for AVT03 and Prolia.
Maximum serum concentration Cmax from day 0 to day 252 | Day 1(week 1) to Day 252 (week 36)
  Venous blood samples will be collected for measurement of maximum serum concentration (Cmax) of AVT03 and Prolia.

SECONDARY OUTCOMES:
PD_AUCE0 for CTX-1 (% inhibition) | Day 1(week 1) to Day 252 (week 36)
  Venous blood samples will be collected for measurement of serum concentration of AVT03 and Prolia
PK area under the concentration-time curve (AUC0-24) from Day 0 to Day 252 | Day 1(week 1) to Day 162 (week 24)]
  Venous blood samples will be collected for measurement of serum concentration of AVT03 and Prolia
Safety incidence, nature and severity of adverse events | Screening to Day 252 (week 36)
Immunogenicity presence and titers of ADAs and presence of nAbs against AVT03 and Prolia | Time Frame: Day 1(week 1) to Day 252 (week 36)
  Venous blood samples will be collected for measurement of antidrug-antibodies against of AVT03 and Prolia

CONTACTS AND LOCATIONS:
Overall Officials: Felicitas Bullo, Study Director — Alvotech
Locations (4):
- Nucleus Network, Herston, Australia
- New Zealand (2):
  - NZCR Christchurch, Christchurch, Christchuch
  - NZCR Auckland, Auckland
- Farmovs, Bloemfontein, South Africa

REFERENCES:
- [Derived] Pretorius A, Bullo F, Jaskiewicz L, Stamatakos S, Otto H, Rai M, Ruffieux R, Sattar A, Leutz S, Berti F. A randomized, double-blind, single dose, parallel group, 2-arm study assessing the pharmacokinetic similarity, pharmacodynamic, safety, tolerability, and immunogenicity profiles of biosimilar candidate AVT03 (60 mg/mL) in healthy male adults. Expert Opin Investig Drugs. 2025 Jun;34(6):527-537. doi: 10.1080/13543784.2025.2505466. Epub 2025 May 16. PMID 40357744